CLINICAL TRIAL: NCT06265636
Title: Transcutaneous Mandibular Nerve Electrical Stimulation for the Management of Pain and Function in Patients With Temporomandibular Disorders
Brief Title: Electrical Stimulation of the Mandibular Nerve for Pain and Function Management in Temporomandibular Disorders
Acronym: Origenkine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OrigenKinesis fisioterapia (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Hector Mardomingo Medialdea, Director, OrigenKinesis fisioterapia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006202325523
Record Dates: First submitted 2024-01-16; First posted 2024-02-20 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Transcutaneous Electric Nerve Stimulation; Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Intervention Model Description: Subjects who participate in the study will receive, in the case of the experimental group, 10 minutes of manual therapy and exercises and 10 minutes of percutaneous electrical nerve stimulation (PENS) guided by ultrasound. In the case of the control group, they will receive 20 minutes of manual therapy and exercises. The treatment will consist of one session per week for three weeks (a total of 3 sessions). Each session will last 30 minutes, of which 10 minutes will be used for the initial evaluation and 20 minutes for the assigned treatment. Two weeks after the last session, a final evaluation without treatment will be performed.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Manual Therapy, exercise and percutaneous electrical nerve stimulation.
  Interventions: Procedure: Percutaneous nerve stimulation; Other: Manual therapy; Other: exercise
- Control Group (Active Comparator): Manual Therapy, exercise.
  Interventions: Other: Manual therapy; Other: exercise

INTERVENTIONS:
Procedure: Percutaneous nerve stimulation — Percutaneous nerve stimulation (PENS) involves inserting a dry needling needle through muscle tissue until it reaches a nerve branch. At this point, a bipolar TENS current with different parameters is applied to the needle with the goal of improving the patient's pain perception.
  Other Names: PENS
  Arms: Experimental Group
Other: Manual therapy — Digital pressure techniques in muscle areas with the aim of reducing the perception of stiffness and pain
Other: exercise — Exercises for improving mandibular mobility, occlusion coordination and regulation of temporomandibular muscle tone

SUMMARY:
Temporomandibular disorders (TMD) encompass dysfunction and pain of the masticatory muscles and temporomandibular joint (TMJ). Pain in the TMJ, restricted jaw movement, and joint sounds are common conditions in this disorder. This can impact patients' ability to perform daily activities such as eating, speaking, laughing, or yawning, significantly affecting their quality of life.

The TMJ and masticatory muscles are innervated by the auriculotemporal branch and the mandibular nerve (V3), a branch of the trigeminal nerve. An estimated 60% to 70% of the population shows signs of TMD, of which up to 12% report intense symptoms requiring treatment.

Percutaneous electrical nerve stimulation (PENS) could be a clinically relevant therapy in TMD patients applied through minimally invasive physiotherapy. To our knowledge, there are no trials evaluating the non-surgical clinical efficacy of PENS on the mandibular nerve.

The project's objective is to assess the effectiveness of PENS on the mandibular nerve in this type of condition.

DETAILED DESCRIPTION:
Pain is the most common and limiting feature of Temporomandibular Disorders (TMD), affecting approximately 75% of the population at some point in life. These disorders involve dysfunction and pain in the masticatory muscles and temporomandibular joint, impacting patients' quality of life. An estimated 60-70% of the population shows signs of TMD, with up to 12% requiring treatment. The peak incidence occurs between 20 and 40 years, predominantly affecting women (8:1 compared to men).

Temporomandibular Disorder often coexists with other medical conditions, such as headaches. The most common diagnoses are myofascial pain, followed by disc displacement with reduction and arthralgia. Prevalence ranges from 3% to 15%, with new case rates between 2% and 4%. Prognosis for myofascial TMD varies, with studies indicating persistence, remission, and relapse.

The economic cost associated with TMD is significant, with studies revealing considerable expenses on treatments. The multifactorial pathophysiology of myofascial pain is influenced by bruxism, stress, psychological conditions, and fibromyalgia. Risk factors include genetics, psychological stress, and parafunctional habits. Clinical manifestations include pain, decreased jaw mobility, and additional symptoms in the head and neck. Diagnosis involves physical examination, palpation of muscles and joints, and imaging tests such as magnetic resonance imaging. Specific diagnostic criteria have been proposed.

Conservative treatment, including physiotherapy, manual therapy, exercises, splints, and pharmacological modalities, is the primary option. However, there are limitations in the effectiveness of some approaches. Physiotherapy is considered effective by 72% of respondents in the United Kingdom.

The musculoskeletal system related to the temporomandibular joint (TMJ) consists of masticatory, facial expression, and neck muscles, playing specific roles in jaw movement. Elevator muscles (masseter, temporal, and medial pterygoid) close the mouth, depressors (digastric and lateral pterygoid) open it, protractors (temporal and lateral pterygoid) move it forward, and retractors (masseter and medial pterygoid) move it backward. Facial expression and neck muscles contribute to additional functions.

Motor innervation of the TMJ comes from the trigeminal nerve, specifically its mandibular branch (V3), which also innervates masticatory muscles. This nerve divides into branches such as the ophthalmic, maxillary, and mandibular, providing sensitivity to different areas of the face, mouth, and jaw.

Blood supply to the TMJ occurs through the superficial temporal artery and the mandibular artery, supplying blood to the skin, muscles, and surrounding joint structures.

Regarding the biomechanics and functionality of the TMJ, its complexity and crucial role in jaw movements such as chewing, speaking, and yawning are emphasized.

Manual therapy, specifically cervico-mandibular therapy, has shown significant improvements in disability related to temporomandibular disorders (TMD). The combination of manual therapy for the orofacial region and the cervical spine has proven to be more effective than home exercises or cervical treatment alone.

Therapeutic exercise in the TMJ has demonstrated moderate short-term effects and variable long-term effects in reducing pain and improving range of motion in patients with TMJ dysfunction. Passive and active stretches, as well as postural exercises, are useful for increasing range of motion and reducing pain.

Percutaneous electrical nerve stimulation (PENS) emerges as a relevant option for managing pain in TMD patients. PENS, applied through ultrasound-guided needles, can influence orofacial pain and jaw movement, offering analgesic benefits through peripheral and central mechanisms. PENS is considered a minimally invasive intervention and has been successfully used in chronic pain treatment.

In summary, a detailed understanding of the anatomy, function, innervation, and vascularization of the TMJ, combined with therapeutic approaches such as manual therapy, exercise, and PENS, is essential for comprehending and effectively addressing temporomandibular disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients with local myofascial pain and/or increased tension in the masticatory muscles.
* Patients with myofascial pain from temporomandibular disorder (TMD) at the time, diagnosed according to the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD).
* Absence of temporomandibular disc displacement with or without reduction.
* Pain in the masticatory muscles associated with limited mouth opening (<40mm).
* Good general health (absence of chronic diseases that may affect the temporomandibular joint or masticatory muscles).
* Written consent to participate in the study.

Exclusion Criteria:

* Injury to the face or head during the research participation.
* Undergone surgical procedures performed in the craniocervical region and degenerative neurological diseases.
* Sudden illness of the patient that prevented participation in the study.
* Will to end participation in the study.
* Less than 2 weeks of evolution.
* Inability to understand instructions or sign the informed consent.
* Minor patients.
* Regular medication, such as muscle relaxants, anticonvulsants, antidepressants, or anxiolytics
* Facial paralysis.
* Presenting a disease or infectious/inflammatory process of dental origin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-17 (Actual); Primary Completion 2027-01-20 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
pain intensity | At the beginning of each intervention session and one month after the end of the last intervention.
  Numerical Pain Rating Scale (NPRS) (Appendix 2). Pain at rest and with chewing on a visual analogue scale. The minimum value is 0, and the maximum is 10. Higher values indicate more pain.
Pressure pain thresholds (PPT) | At the beginning of each intervention session and one month after the end of the last intervention.
  A pressure algometer (kg/cm2) will be used. The measurement will be taken with which the minimum amount of pressure applied to the masseter muscle produces pain.
Pain-free mandibular opening range of motion | At the beginning of each intervention session and one month after the end of the last intervention.
  herabite® System ruler (Appendix 3). 6 mm has been determined as the minimum detectable change in maximum mouth opening [56]. Mandibular range of motion (maximum mouth opening) will be measured with a device that allows the evaluation of mouth movements in millimeters.

SECONDARY OUTCOMES:
Self-reported quality of life (SF-12) | At the beginning of the first intervention and one month after the last intervention.
  The SF-12 Life Satisfaction Scale measures health-related quality of life. While not directly scoring life satisfaction, it assesses physical and mental health perceptions. Scores for each dimension provide insights into overall life satisfaction. The SF-12 comprises 12 questions across 8 dimensions, such as physical limitations, social roles, pain, and mental health. These yield two summary components: Physical Component Summary (PCS) and Mental Component Summary (MCS). Scores, standardized with a mean of 50 and a standard deviation of 10 in the general population, indicate better health-related quality of life with higher scores.
Electromyographic activation rate of the masseter muscle. | At the beginning of the first intervention and one month after the last intervention.
  The surface EMG recording will be obtained using an 11 mDurance® four-channel surface electromyograph. The unit of measurement will be in picovolts. Higher picovolt detection indicates greater muscle excitability. Visual graphs will be used to represent the amount of activation of the masseter muscle. The EMG signal was captured in two tasks: during resting mandibular position (MR) and during a 5-second sustained maximum occlusion contraction (MVC).

CONTACTS AND LOCATIONS:
Locations (1):
- Origenkinesis Fisioterapia, Alcorcón, Madrid, Spain

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT06265636/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT06265636/ICF_001.pdf